CLINICAL TRIAL: NCT01840397
Title: Elevated Levels of S-100B and Neuron-specific Enolase (NSE) in Spine Surgery: A Comparison of Serum Levels With Surgery for Long-bone Fractures
Brief Title: Neuromarker S-100B as Diagnostic Tool
Acronym: SpineSurgery
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Harald Wolf, MD, Dr. Harald Wolf, Medical University of Vienna
Other Study IDs: Wolf-6
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Spinal Injury
Keywords: S-100B; NSE
MeSH Terms: conditions — Spinal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum levels of the biomarkers S-100B and NSE are measured
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spine surgery: Patients undergoing spine surgery
- Bone surgery: Patients undergoing bone surgery for fracture treatment other than spine fractures

SUMMARY:
The hypothesis of this study is to find evidence if there is an influence of spine surgery on the serum levels of two proteins secreted from neuronal cells.

DETAILED DESCRIPTION:
The question, if there is an effect on the cerebrospinal system during spine surgery, which can be traced by monitoring serum levels of neuromarkers is not yet answered. This study has its background from other studies on patients with traumatic brain injury (TBI), in whom elevated serum levels of the two neuromarkers S-100B and NSE are associated with injury severity, neuronal damage, brain, tissue damage, and outcome. Patients undergoing spine surgery with or without pre-existing traumatic neurologic symptoms are planned to be the study cohort. Pre- and postoperatively the serum levels of S-100B and NSE are obtained and are statistically compared with patients undergoing other types of bone-related surgery.

ELIGIBILITY:
Inclusion Criteria:

* spine fracture

Exclusion Criteria:

* additional traumatic brain injury
* fractures of the long bones
* polytrauma
* severely injured patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spine fractures undergoing spine surgery for fracture stabilization
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
S-100B levels | 4 hours
  average timeframe between blood withdrawal (twice, pre-and post-operatively)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Wolf, M.D., Principal Investigator — Medical University of Vienna, Department for Trauma Surgery
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Cao F, Yang XF, Liu WG, Hu WW, Li G, Zheng XJ, Shen F, Zhao XQ, Lv ST. Elevation of neuron-specific enolase and S-100beta protein level in experimental acute spinal cord injury. J Clin Neurosci. 2008 May;15(5):541-4. doi: 10.1016/j.jocn.2007.05.014. Epub 2008 Mar 14. PMID 18343116
- [Background] Marquardt G, Setzer M, Theisen A, Tews DS, Seifert V. Experimental subacute spinal cord compression: correlation of serial S100B and NSE serum measurements, histopathological changes, and outcome. Neurol Res. 2011 May;33(4):421-6. doi: 10.1179/1743132810Y.0000000005. PMID 21535942
- [Background] Marquardt G, Setzer M, Szelenyi A, Seifert V, Gerlach R. Prognostic relevance of serial S100b and NSE serum measurements in patients with spinal intradural lesions. Neurol Res. 2009 Apr;31(3):265-9. doi: 10.1179/174313209X382287. Epub 2008 Nov 26. PMID 19040802